CLINICAL TRIAL: NCT03177148
Title: Population Effects of Motivational Interviewing on Pediatric Obesity in Primary Care
Brief Title: Population Effects of MI on Pediatric Obesity in Primary Care
Acronym: BMi2+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Academy of Pediatrics (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ken Resnicow, Professor, Health Behavior & Health Education, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BMi2+; 5R01HL128231-05 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: After two years of intervention arm study, the usual care arm will receive MI training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): * 1-2 pediatric clinicians per practice will be trained in study procedures, current obesity treatment guidelines, and obesity billing and coding via telephone and webinar
  * NO active enrollment of parents
  * Secure extraction of HIPAA limited Electronic Health Record (EHR) and billing data from practices for outcomes analyses
  At the end of the intervention period, 1-2 pediatric clinicians will be offered the in-person MI training and DVD materials
  Interventions: Behavioral: Usual Care
- Intervention by Clinicians (Experimental): * Pediatric Clinicians complete surveys during enrollment and end of the intervention
  * 1-2 clinicians from each practice will receive 2.5 days of in-person MI training, two scored encounters with a standardized patient, and an interactive DVD MI booster training system focusing on pediatric obesity.
  * Enroll 35 eligible parents per practice
  * Clinicians give up to 4 in-person, MI sessions to enrolled parents over 2 years.
  Dietitians will provide up to 6 telephone counseling sessions.
  •Parents will complete surveys after enrollment and at the end of intervention
  Interventions: Behavioral: Intervention by Clinicians

INTERVENTIONS:
Behavioral: Intervention by Clinicians — •Parents will complete surveys after enrollment and at the end of intervention and participate in intervention visits by pediatric clinicians and telephonic counseling with Registered Dietitians (RDs).
  Intervention by pediatric clinicians: up to 4 sessions of MI, in-person Intervention by RDs: up to 6 sessions of MI via telephone.
  Other Names: MI Intervention
  Arms: Intervention by Clinicians
Behavioral: Usual Care — Pediatric clinicians provide care as normal
  Arms: Usual Care

SUMMARY:
In this cluster randomized effectiveness trial, pediatric primary care practices will be recruited from the American Academy of Pediatrics' national Pediatric Research in Office Settings (PROS) practice-based research network, as well as the client database of the Physician's Computer Company (PCC) - an Electronic Health Record (EHR) vendor. We will recruit 18 practices. 9 practices will be randomized to the Intervention arm and 9 practices to Usual Care. Intervention arm practices will select 1-2 pediatric clinicians, including pediatricians (PED) and nurse practitioners (NP), to receive in-person training in Motivational Interviewing (MI), behavioral therapy, billing and coding, and study procedures. Usual Care practices will select 1-2 pediatric clinicians to receive billing / coding and study protocol training only, via telephone and webinar; they will be offered in-person MI training at the close of the trial. Around 316 parents of overweight or obese children (BMI > 85th percentile for age and gender) between 3 and 11 years of age at baseline that are patients of participating Intervention arm clinicians will be enrolled. Over 24 months, these parents may receive up to 4 in-person, MI-based counseling sessions with a trained pediatric clinician and up to 6 telephone counseling sessions with an MI-trained Registered Dietician (RD). There will be no study-specific contact with parents or their children in Usual Care practices during the trial - they will continue to receive usual care. EHR and billing data for all 3-11 year old children within all participating practices will be extracted by PCC to permit determination of the effectiveness of the intervention versus usual care on change in BMI z-score among 3 groups: 1) all eligible children in the Intervention arm), 2) all eligible children whose parent actively participates in the trial , and 3) all 3-11 year old children in all participating practices.

ELIGIBILITY:
Inclusion Criteria:

* For Practices: Currently use Physician's Computer Company (PCC) as their Electronic Health Record (EHR) vendor
* For Clinicians: Have been employed by the practice for at least 1 year on or before July 1, 2017 Work > half time (at least 6 sessions per week)
* For Parents: Parent or legal guardian of a child that meets the following criteria: At least 3 but not yet 12 years of age on the date of the baseline data pull (estimated to occur in the summer or fall of 2017). BMI for age and gender > 85th percentile - documented at an office visit that occurred during the 12 months prior to the baseline data pull. Most recent well-child visit was with a participating study clinician during the 24 months prior to the baseline data pull

Exclusion Criteria:

* For Practices: Offer a comprehensive weight loss program or access to a RD at or through the practice. Unable or unwilling to send all participating study clinicians to in-person training.Unable or unwilling to identify and assign a study coordinator for the study
* For Clinicians: > 1 day of prior training in MI within the past 10 years. Prior participation in the AAP/PROS Healthy Lifestyles Pilot Study (HLS; AAP IRB protocol # 01SC01) or Brief Motivational Interviewing to Reduce Body Mass Index (BMI2) Study (AAP IRB protocol # 07RE01).
* For Parents: Does not speak either English or Spanish. Parent or legal guardian of a child who has any of the following documented in their EHR: Type I or Type II diabetes. Daily or chronic use of medications known to affect growth and mood / behavior (growth hormones, SSRIs, stimulants).Use of atypical antipsychotics. A chronic, limiting, severe medical disorder, syndrome, or other condition (e.g., Downs syndrome, cerebral palsy)

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 352 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Resnicow, Ph.D., Principal Investigator — University of Michigan; Emerson Delacroix, M.A.C.P., Study Director — University of Michigan
Locations (1):
- Pediatric Research in Office Settings, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
An external DSMB will be used. They will meet at least once a year, and will convene as needed to review potential adverse events.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study teams at University of Michigan and the American Academy of Pediatrics disseminate the protocol with any deviations or adverse events to the external DSMB for their annual meeting, and at the conclusion of the study. Data will be de-identified after the intervention phase ends which is planned for May 2021.
Access Criteria: DSMB members and study team members have access to the data and results of the study.

REFERENCES:
- [Derived] Wright ME, Delacroix E, Sonneville KR, Considine S, Proctor T, Steffes J, Harris D, Shone LP, Woo H, Vaughan R, Grundmeier RW, Fiks AG, Stockwell MS, Resnicow K. Reducing paediatric overweight and obesity through motivational interviewing: study protocol for a randomised controlled trial in the AAP PROS research network. BMJ Open. 2020 Jul 28;10(7):e035720. doi: 10.1136/bmjopen-2019-035720. PMID 32723736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Practices and pediatric clinicians were recruited through the AAP Pediatric Research in Office Settings (PROS) network who used Physician's Computer Company (PCC), an EHR vendor tailored to pediatric practices. Pediatric clinicians were enrolled in intervention arm and usual care arm and completed baseline and follow-up surveys.
  Parents/caregivers were only enrolled in the intervention arm and completed baseline and follow-up surveys. Parents chose one of their eligible children to enroll.
Pre-assignment Details: 18 pediatric practices were randomized to the intervention or usual control arm.
  Parents/caregivers were only enrolled in the intervention arm provided self-report survey data.
  Children were enrolled by their Parent/Caregiver in the intervention arm ONLY. Childrens data was extracted from the EHR for BOTH the intervention and usual care arm. NO children were enrolled in the usual care arm, only child BMI data from enrolled pediatric clinicians in the usual care arm were used.
Units Other Than Participants: Pediatric practices
Groups:
- Intervention by Clinicians: * Pediatric Clinicians complete surveys during enrollment and end of the intervention
  * 1-2 clinicians from each practice will receive 2.5 days of in-person MI training, two scored encounters with a standardized patient, and an interactive DVD MI booster training system focusing on pediatric obesity.
  * Enroll 35 eligible parents per practice
  * Clinicians give up to 4 in-person, MI sessions to enrolled parents over 2 years.
  * Dietitians will provide up to 6 telephone counseling sessions.
  * Parents will complete surveys after enrollment and at the end of intervention
- Usual Care: * 1-2 pediatric clinicians per practice will be trained in study procedures, current obesity treatment guidelines, and obesity billing and coding via telephone and webinar.
  * NO active enrollment of parents
  * Secure extraction of HIPAA limited Electronic Health Record (EHR) and billing data from practices for outcomes analyses.
  * At the end of the intervention period, 1-2 pediatric clinicians will be offered the in-person MI training and DVD materials.
Period: Overall Study
Arm/Group | Intervention by Clinicians | Usual Care
Started | 340; 9 Pediatric practices (11 pediatric clinicians enrolled from the 9 intervention practices 329 parents/caregivers consented to enroll their child. The actual child was not enrolled. No child interacted with the study team.) | 12; 9 Pediatric practices (12 pediatric clinicians enrolled from the 9 usual care practices)
Completed | 289; 8 Pediatric practices (Enrolled parent/caregiver provided child BMI data to enrolled pediatric clinician at baseline and follow-up. 1 intervention clinician died during the intervention; their practice and other intervention clinician withdrew from the study.) | 11; 8 Pediatric practices (Children seen by Usual Care arm pediatric clinicians, with BMI data in their EHR at baseline and follow-up, were matched with intervention arm children after the completion of the study. 1 practice ceased using the EHR and had to withdraw from the study.)
Not Completed | 51; 1 Pediatric practices | 1; 1 Pediatric practices
Not completed — Lost to Follow-up | 50 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Parents/caregivers enrolled one child into the intervention. Parents/caregivers completed a baseline survey about the enrolled child. BMI values were extracted from the EHR. Parents/caregivers and intervention pediatric clinicians did not report baseline survey responses for baseline analysis population description. No baseline characteristic data was collected for the Usual Care Arm (clinicians, parents or children).
Arm/Group | Intervention by Clinicians
Number analyzed (Participants) | 329
Age, Categorical [Count of Participants; unit: Participants] — Collected from electronic health record Population: 49 participants could not be contacted for follow-up data
  Participants
    <=18 years | 329
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.93 (2.54)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Collected by survey completed by parent. 67 parents did not complete this baseline survey question leaving 262 as the overall number of baseline participants for this baseline characteristic.
  Participants
    He/Him/His: number analyzed (Participants) | 262
    He/Him/His | 131
    She/Her/Hers: number analyzed (Participants) | 262
    She/Her/Hers | 126
    They/Them/Their: number analyzed (Participants) | 262
    They/Them/Their | 5
Sex: Female, Male [Count of Participants; unit: Participants] — Collected by survey completed by parent. Population: 49 parents did not provide a response to this survey question.
  Participants
    number analyzed (Participants) | 280
    Female | 146
    Male | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 110
  Not Hispanic or Latino | 151
  Unknown or Not Reported | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 52
  White | 161
  More than one race | 34
  Unknown or Not Reported | 67
Region of Enrollment [Count of Participants; unit: Participants] — Population: 49 parents did not provide a response to this survey question leaving 280 as the overall number of participants analyzed for this for baseline characteristic.
  Participants
    United States: number analyzed (Participants) | 280
    United States | 280
Two-level Baseline Body Mass Index Categorical Variable [Count of Participants; unit: Participants]
  Low Baseline BMI (Percentile < 120) | 236
  High Baseline BMI (Percentile >= 120) | 44
  Unknown/Missing | 49

OUTCOME MEASURES:

1. Primary Outcome: Percent Distance From the Sex-age Specific 95th Percentile
Description: Differences between intervention and usual care youth at baseline for distance from the 95th percentile for BMI. BMI data from children seen by Usual Care arm pediatric clinicians were matched (3 to 1) to intervention arm children.
Time Frame: Baseline
Population: Treatment by time interaction predicted distance above the 95th percentile. The Overall Number of Participants Analyzed reflects data extracted from EHR of children who were seen by the enrolled physicians. The overall number of participants analyzed in the usual care arm represents the BMI data extracted from children seen by the enrolled usual care arm clinicians. These children were not considered enrolled.
Measure: Mean (Standard Deviation); unit: % distance from 95th percentile
Groups:
- Usual Care: * 1-2 pediatric clinicians per practice will be trained in study procedures, current obesity treatment guidelines, and obesity billing and coding via telephone and webinar.
  * NO active enrollment of parents and children
  * Secure extraction of HIPAA limited Electronic Health Record (EHR) and billing data from practices for outcomes analyses.
  * At the end of the intervention period, 1-2 pediatric clinicians will be offered the in-person MI training and DVD materials.
  * BMI data from children seen by Usual Care arm pediatric clinicians were reviewed and the BMI data in the EHR at baseline and follow up were matched with the intervention arm children after the study.
Arm/Group | Intervention by Clinicians | Usual Care
Number analyzed (Participants) | 280 | 840
% distance from 95th percentile | 106.4 (15.88) | 102.7 (13.32)

2. Secondary Outcome: Raw BMI Score
Description: Differences between intervention and usual care youth at baseline for raw BMI score
Time Frame: Baseline
Population: 3:1 matched cohort. The Overall Number of Participants Analyzed reflects data extracted from EHR of children who were seen by the enrolled physicians. The overall number of participants analyzed in the usual care arm represents the BMI data extracted from children seen by the enrolled usual care arm clinicians. These children were not considered enrolled.
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Usual Care: * 1-2 pediatric clinicians per practice will be trained in study procedures, current obesity treatment guidelines, and obesity billing and coding via telephone and webinar.
  * NO active enrollment of parents and children
  * Secure extraction of HIPAA limited Electronic Health Record (EHR) and billing data from practices for outcomes analyses.
  * At the end of the intervention period, 1-2 pediatric clinicians will be offered the in-person MI training and DVD materials.
Arm/Group | Intervention by Clinicians | Usual Care
Number analyzed (Participants) | 280 | 840
kg/m^2 | 21.4 (4.39) | 20.5 (3.51)

ADVERSE EVENTS:
Time Frame: 4-years
Description: Only the intervention arm was assessed for adverse events. Adverse events were not monitored/assessed in the parent/caregiver populations; only children were monitored/assessed for adverse events
Groups:
- Intervention Clinicians; Intervention Parents/Caregivers; Intervention Children: * Pediatric Clinicians complete surveys during enrollment and end of the intervention
  * 1-2 clinicians from each practice will receive 2.5 days of in-person MI training, two scored encounters with a standardized patient, and an interactive DVD MI booster training system focusing on pediatric obesity.
  * Enroll 35 eligible parents per practice
  * Clinicians give up to 4 in-person, MI sessions to enrolled parents over 2 years.
  * Dietitians will provide up to 6 telephone counseling sessions.
  * Parents will complete surveys after enrollment and at the end of intervention
Arm/Group | Intervention Clinicians | Intervention Parents/Caregivers | Intervention Children
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/0 | 0/329
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/0 | 0/329
Other Adverse Events (participants affected / at risk) | 0/11 | 0/0 | 1/329
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Clinicians (N=11) | Intervention Parents/Caregivers (N=0) | Intervention Children (N=329)
Other Adverse Event (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT03177148/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03177148/SAP_001.pdf